CLINICAL TRIAL: NCT06844006
Title: Assessment of Digital Care on Clinical Impact and Efficiency Using a Stepped Wedge Cluster RCT in Heart Failure Patients: the ADMINISTER II Trial
Brief Title: Investigating the Impact of Nudging Cardiologists to Prescribe Guideline-directed Medical Therapy in Heart Failure Patients
Acronym: ADMINISTER II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medisch Spectrum Twente (Other)
Collaborators: Onze Lieve Vrouwe Gasthuis (Other); St. Antonius Hospital (Other); Martini Hospital Groningen (Other); Catharina Ziekenhuis Eindhoven (Other); Canisius Wilhelmina Ziekenhuis (CWZ) (Unknown); Maasstad Hospital, Rotterdam (Unknown)
Responsible Party: Principal Investigator, Mark Schuuring, Assistent Professor M.J. Schuuring (M.D., Ph. D., FESC, FEACVI, FHFA), Medisch Spectrum Twente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADMINISTER II
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: Digitial Care; Home monitoring; Heart Failure; Nudging
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Randomized Controlled Trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Other): All cardiologists will be nudged during the trial. with the use of a stepped wedge design there will be a structured embedding in the current standard of care.
  Interventions: Combination Product: Nudging

INTERVENTIONS:
Combination Product: Nudging — Clinicians will be nudged with a prompt, based on remote monitoring data, current medication data, contraindications, in the electronic patient dossier whether further optimization to guideline directed medical therapy (GDMT) is possible.

SUMMARY:
This study investigates the impact of a nudge-based intervention on improving guideline directed medical therapy (GDMT) prescription among cardiologists. Using a stepped wedge randomized controlled trial design, we assess whether digital decision support-leveraging home monitoring and clinical data-enhances adherence to guideline-recommended medication titration. The primary outcomes include HF related hospitalization rates and all cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* All heart failure diagnoses
* >18 years

Exclusion Criteria:

* Not understanding the Dutch Language.
* Allergies that make uptitration impossible.
* Admission to hospice or palliative care.
* Severe psychological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1320 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
HF related hospitalization | From enrollment to the end of the design (15 months).
  The frequency of HF related hospitalization and duration of the hospitalization.
All cause death | All cause death rate during the 15 month duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Man JP, Koole MAC, Meregalli PG, Handoko ML, Stienen S, de Lange FJ, Winter MM, Schijven MP, Kok WEM, Kuipers DI, van der Harst P, Asselbergs FW, Zwinderman AH, Dijkgraaf MGW, Chamuleau SAJ, Schuuring MJ. Digital consults in heart failure care: a randomized controlled trial. Nat Med. 2024 Oct;30(10):2907-2913. doi: 10.1038/s41591-024-03238-6. Epub 2024 Aug 31. PMID 39217271
- See also: Related Info — https://www.nature.com/articles/s41591-024-03238-6